CLINICAL TRIAL: NCT03285230
Title: The French E3N Prospective Cohort Study (Etude Epidémiologique auprès de Femmes de la Mutuelle Générale de l'Education Nationale)
Brief Title: The French E3N Prospective Cohort Study
Acronym: E3N
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Université Paris-Sud (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: C 95-01
Record Dates: First submitted 2017-07-27; First posted 2017-09-15 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer; Colo-rectal Cancer; Parkinson Disease; Asthma; Diabetes; Inflammatory Bowel Diseases; Melanoma; Endometriosis; Thyroid Cancer; Hypertension; Endometrial Cancer; Crohn Disease; Depression; Cardiovascular Diseases
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Parkinson Disease; Asthma; Diabetes Mellitus; Inflammatory Bowel Diseases; Melanoma; Endometriosis; Thyroid Neoplasms; Hypertension; Endometrial Neoplasms; Crohn Disease; Depression; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 25000 blood samples; 47000 saliva samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The French E3N cohort was initiated in 1990 to investigate the risk factors associated with cancer and other major non-communicable diseases in women.

The participants were insured through a national health system that primarily covered teachers, and were enrolled from 1990 after returning baseline self-administered questionnaires and providing informed consent. The cohort comprised nearly 100 000 women with baseline ages ranging from 40 to 65 years.

Follow-up questionnaires were sent approximately every 2-3 years after the baseline and addressed general and lifestyle characteristics together with medical events (cancer, cardiovascular diseases, diabetes, depression, fractures and asthma, among others). The follow-up questionnaire response rate remained stable at approximately 80%.

A biological material bank was generated and included blood samples collected from 25 000 women and saliva samples from an additional 47 000 women.

Ageing among the E3N cohort provided the opportunity to investigate factors related to agerelated diseases and conditions as well as disease survival.

DETAILED DESCRIPTION:
Who is in the cohort? In June 1990, a questionnaire was sent to 500 000 women who had been born between 1925 and 1950 and were insured by the Mutuelle Générale de l'Education Nationale (MGEN), a national health insurance plan that primarily covers teachers. The questionnaire was sent along with a leaflet explaining that an Inserm research team was launching a study of cancer risk factors and that participation would require filling in questionnaires every 2-3 years as well as the submission of a signed consent form providing permission to obtain information about each participant's vital status, address changes and medical expense reimbursements from the insurance plan. Nearly 100 000 women volunteered.

How often have they been followed-up? Until now, nine follow-up questionnaires have been sent every 2-3 years from the baseline. Approximately half of the answers were obtained after the first mailing. Two reminders were sent thereafter. The questionnaires were accompanied with newsletters that informed participants about the major results obtained to date. The participation rate remained high (77-92% according to the questionnaires) and the lost to follow-up rate was minimal because of the ability to trace non-respondents through their insurance plan files. The questionnaires were accurately filled in, with few missing or unacceptable answers.

What has been measured? To date, 11 self-administered questionnaires have been sent. The collected data are sociodemographic factors, anthropometric measurements, reproductive factors, hormonal treatments, health behaviour and lifestyle. Each follow-up questionnaire also recorded the participant's health status. The questionnaires are available at www.e3n.fr .

The questionnaires are anonymous and identified with an identification number and pin code that can be rapidly scanned to identify the respondents. The questionnaires are optically scanned and all answers are checked on screen. The scanned images are saved to allow data entry at a later time, including information regarding the addresses of medical doctors (18 000 to date) or drug names (pre-listed to avoid errors). The longitudinal data (repeats of identical questions for the purpose of updating information about topics such as menopause or smoking) are routinely homogenized. Several validation studies (e.g. dietary and anthropometrical data studies) have been performed and have revealed very satisfactory results.

Self-reported cases of cancer are validated and coded after reviewing the pathology reports obtained from medical practitioners, and nearly 90% of all cancer cases are histologically confirmed. Other diseases are also validated (e.g. diabetes, myocardial infarction, stroke, Parkinson disease) by requesting additional information about the participants (e.g. glycosylated haemoglobin levels, fracture-related circumstances, drug names) and sending questionnaires to medical doctors.

Additionally, a biological material bank was generated. Blood samples were initially collected from 1994-99. The participation rate among the invited participants was approximately 40%; this yielded approximately 25 000 blood samples that were each separated into 28 aliquots (e.g. plasma, serum, leukocytes, erythrocytes). Plastic straws were used to store each participant's samples in liquid nitrogen containers. The bio-repositories are located at the IARC (Lyon) and the EFS (Etablissement Français du Sang, Annemasse). Since 2004, approximately 10 case-control studies have been conducted (approximately 1 800 cases and 3 500 controls) with regard to the measurements of various biomarkers (e.g. fatty acids, calcium, vitamin D, vitamin B, cholesterol and C-reactive protein). A metabolomics study is currently ongoing.

From 2009-11, saliva samples (Oragene, DNA Genotek, Kanata, ON, Canada) were requested from 68 242 living women and were obtained from 47 000 women (participation rate, 69%). Salivary DNA has been extracted and has been used for genotyping in two case-control studies (approximately 2 500 cases and 850 controls) since December 2010.

The research team is currently planning to set up a tumour tissue bank and will begin with the collection of breast cancer tissues.

What has it found? The E3N cohort has produced a spectrum of results regarding the complex roles played by nutrition, hormonal factors, physical activity, anthropometric characteristics and other major lifestyle-related factors with respect to various diseases.

ELIGIBILITY:
Inclusion Criteria:

* only women
* born between 1925 and 1950
* insured by the Mutuelle Générale de l'Education Nationale (MGEN)

Exclusion Criteria:

- men

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort comprised nearly 100 000 women with baseline ages ranging from 40 to 65 years, all insured through a French national health system (MGEN).
Sampling Method: Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 1990-06-15 (Actual); Primary Completion 1991-11-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements | From 1990 until now
  Height, weight, hip circumference and waist circumference
Educational level | 1990
Professional activity | 1992 and 2005
  Insee categories
Age at cessation of activity | From 2005 until now
Menstrual factors | From 1990 to 2002
  Age at menarche, length of menstrual cycle
Reproductive history | From 1990 to 1992
  Number of pregnancies, age at each pregnancy, durations and outcomes of pregnancies, breastfeeding, infertility
Menopause | 1990, 1995, 1997, 2000, 2002, 2005
  Age, type
Hormonal Treatments | From 1992 to 2008
  Menopausal Hormonal Treatments (MHT), oral contraceptives
Tobacco consumption | From 1990 until now
  Type, quantity, time of smoking
Alcohol consumption | 1993, 1997, 2005
  Type of alcohol, quantity
Physical activity | 1990,1997,2002, 2005, 2014
  Moderate and intense activity, sedentarity
Diet questionnaire | 1993 and 2002
  Precise annual diet questionnaire
Family history of diseases | 1990 to 2005
  Cancer, diabetes and cardiovascular diseases
Medication use | From 1990 until now
  linked with the drug reimbursement files from the health insurance
Medical and surgical history | From 1990 until now
Mental Health | From 1990 until now
  Centre for Epidemiologic Studies Depression Scale (CESD) and Depression
Health outcomes | From 1990 until now

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Severi, PhD, Study Director — INSERM (Institut National de la Sante et de la Recherche Medicale); Marie-Christine Boutron-Ruault, PhD, Principal Investigator — INSERM (Institut National de la Sante et de la Recherche Medicale)

REFERENCES:
- [Background] Clavel-Chapelon F; E3N Study Group. Cohort Profile: The French E3N Cohort Study. Int J Epidemiol. 2015 Jun;44(3):801-9. doi: 10.1093/ije/dyu184. Epub 2014 Sep 10. PMID 25212479
- [Derived] Dusser P, Nguyen Y, Perrin C, Frenoy P, Mariette X, Boutron-Ruault MC, Varraso R, Severi G, Salliot C, Seror R. Early-life animal and farming exposures and the risk of rheumatoid arthritis: findings from the E3N French cohort study. RMD Open. 2025 Dec 7;11(4):e005954. doi: 10.1136/rmdopen-2025-005954. PMID 41360603
- [Derived] Auguste A, Jansana A, Freisling H, Ferrari P, Laouali N, Severi G, Kvaskoff M. Impact of Hypertension on Cancer Stage at Diagnosis Among French Women: The E3N Prospective Cohort. Cancer Med. 2025 Aug;14(15):e71021. doi: 10.1002/cam4.71021. PMID 40719276
- [Derived] Klu YE, Amazouz H, Canonico M, Guenel P, Kvaskoff M, Severi G, Radoi L, Auguste A. Association Between Hormonal Factors and Risk of Lung and Upper Aerodigestive Tract Cancer in French Women: The E3N Prospective Cohort Study. Cancer Rep (Hoboken). 2025 Jun;8(6):e70223. doi: 10.1002/cnr2.70223. PMID 40490966
- [Derived] Koemel NA, Shah S, Senior AM, Severi G, Mancini FR, Gill TP, Simpson SJ, Raubenheimer D, Boutron-Ruault MC, Laouali N, Skilton MR. Macronutrient composition of plant-based diets and breast cancer risk: the E3N prospective cohort study. Eur J Nutr. 2024 Aug;63(5):1771-1781. doi: 10.1007/s00394-024-03379-x. Epub 2024 Apr 18. PMID 38635026
- [Derived] Shah S, Mahamat-Saleh Y, Ait-Hadad W, Koemel NA, Varraso R, Boutron-Ruault MC, Laouali N. Long-term adherence to healthful and unhealthful plant-based diets and breast cancer risk overall and by hormone receptor and histologic subtypes among postmenopausal females. Am J Clin Nutr. 2023 Mar;117(3):467-476. doi: 10.1016/j.ajcnut.2022.11.019. PMID 36872016
- [Derived] Shah S, Mahamat-Saleh Y, Hajji-Louati M, Correia E, Oulhote Y, Boutron-Ruault MC, Laouali N. Palaeolithic diet score and risk of breast cancer among postmenopausal women overall and by hormone receptor and histologic subtypes. Eur J Clin Nutr. 2023 May;77(5):596-602. doi: 10.1038/s41430-023-01267-x. Epub 2023 Feb 1. PMID 36726032
- [Derived] Frenoy P, Perduca V, Cano-Sancho G, Antignac JP, Severi G, Mancini FR. Application of two statistical approaches (Bayesian Kernel Machine Regression and Principal Component Regression) to assess breast cancer risk in association to exposure to mixtures of brominated flame retardants and per- and polyfluorinated alkylated substances in the E3N cohort. Environ Health. 2022 Feb 26;21(1):27. doi: 10.1186/s12940-022-00840-4. PMID 35216589
- [Derived] Madika AL, MacDonald CJ, Gelot A, Hitier S, Mounier-Vehier C, Beraud G, Kvaskoff M, Boutron-Ruault MC, Bonnet F. Hysterectomy, non-malignant gynecological diseases, and the risk of incident hypertension: The E3N prospective cohort. Maturitas. 2021 Aug;150:22-29. doi: 10.1016/j.maturitas.2021.06.001. Epub 2021 Jun 12. PMID 34274072
- [Derived] Laouali N, Shah S, MacDonald CJ, Mahamat-Saleh Y, El Fatouhi D, Mancini F, Fagherazzi G, Boutron-Ruault MC. BMI in the Associations of Plant-Based Diets with Type 2 Diabetes and Hypertension Risks in Women: The E3N Prospective Cohort Study. J Nutr. 2021 Sep 4;151(9):2731-2740. doi: 10.1093/jn/nxab158. PMID 34236437
- [Derived] Cairat M, Al Rahmoun M, Gunter MJ, Severi G, Dossus L, Fournier A. Antiplatelet Drug Use and Breast Cancer Risk in a Prospective Cohort of Postmenopausal Women. Cancer Epidemiol Biomarkers Prev. 2021 Apr;30(4):643-652. doi: 10.1158/1055-9965.EPI-20-1292. Epub 2021 Feb 2. PMID 33531438
- [Derived] Azevedo Da Silva M, Fournier A, Boutron-Ruault MC, Balkau B, Bonnet F, Nabi H, Fagherazzi G. Increased risk of type 2 diabetes in antidepressant users: evidence from a 6-year longitudinal study in the E3N cohort. Diabet Med. 2020 Nov;37(11):1866-1873. doi: 10.1111/dme.14345. Epub 2020 Jul 2. PMID 32542873
- [Derived] Mahamat-Saleh Y, Cervenka I, Al Rahmoun M, Savoye I, Mancini FR, Trichopoulou A, Boutron-Ruault MC, Kvaskoff M. Mediterranean dietary pattern and skin cancer risk: A prospective cohort study in French women. Am J Clin Nutr. 2019 Oct 1;110(4):993-1002. doi: 10.1093/ajcn/nqz173. PMID 31380561
- See also: website of the study — http://www.e3n.fr